CLINICAL TRIAL: NCT01557751
Title: Preliminary Studies for Whole Genome Association Study (WGAS) in Acute Perioperative Pain
Brief Title: Acute Pain Genomic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Jacques E. Chelly, Professor of Anesthesiology (with Tenure) and Orthopedic Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO09050171; N08PC10039 (Other Grant/Funding Number: US NIH/NIDCR); 1406-0408-CT-20481 (Other Grant/Funding Number: US NIH/NIDCR)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis; Postoperative Pain
Keywords: Total knee arthroplasty; Total knee replacement; Genetics of pain
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Total knee arthroplasty subjects who are genotyped (Other): All patients will have whole blood drawn for genotyping, and participate in the various assessments (psychosocial questionnaires, qualitative sensory testing, etc).
  Interventions: Genetic: Whole blood for genotyping

INTERVENTIONS:
Genetic: Whole blood for genotyping — This study requires genotyping by extracting DNA from blood sample. A blood sample will be drawn once during visit 2 (day of surgery) or any other time prior to that after the signing of informed consent. Four vacutainers of which hold 8.5 mL will be drawn during this time totaling approximately 34 mL of blood which completes the genomic sampling portion of the study.

SUMMARY:
In preparation for future large-scale genome wide association studies, reliable methods must be developed for measuring perceived pain and for estimating the effects of potentially confounding factors such as appropriate covariates. The major objectives of our pilot investigation are to develop optimal methods to characterize the primary endpoint of the study-knee pain, and to gather preliminary data on genetic markers in the human genome that are associated with a certain pain phenotype. The specific issues for this study will be to carry out a preliminary gene association analysis of acute perioperative pain in individuals undergoing total knee replacement and to define a pain phenotype that is composed of multidimensional domains such as opioid consumption, inflammatory markers, anxiety level, degree of catastrophizing, etc. This pain phenotype has to be sensitive enough to pick up changes in pain experience that can be attributed to single nucleotide polymorphisms.

DETAILED DESCRIPTION:
In spite of advances in postoperative management and the standardization of postoperative care, there is a wide variability in the degree of pain relief achieved which cannot be accounted for. The aim of this study is to devise a method for defining a pain phenotype sensitive enough to detect differences in genetic makeup between individuals who undergo a standard surgical procedure (total knee replacement). This methodology will serve as a pilot study for future genome wide association studies. Given the multidimensional aspects of pain experience, the phenotype will be combined of various dimensions comprising postoperative pain. Reports about single nucleotide polymorphisms (SNPs), which account for some of the variability of pain, have been reported in the literature using different pain models. To test the sensitivity of our method of phenotyping, the investigators aim to determine if variability in our clinical phenotypes can be explained by some of the SNPs published in the literature. Patients scheduled for elective unilateral primary total knee arthroplasty will be asked to report on various clinical pain variables, fill psychometric questionnaires, be subjected to quantitative sensory testing, genotyped for a genes associated with pain, and additional SNPs. A composite pain profile will be composed for each patient initially examining five candidate genes and related SNPs to find out the SNPs that are significantly associated with given pain phenotypes. Samples will be banked for future study of other genes associated with pain. Other clinical variables will be collected (e.g. opioid consumption). At six and twelve months, psychological questionnaires and pain questionnaires will be sent to patient. A model using pain during physical therapy as the dependent variable will be fit to the data. Knee joint fluid, urine, and serum will be collected from approximately 30% of the subjects who provide their additional consent cytokine and other inflammatory marker analysis. All biological specimens will be banked for future analysis. This is a pilot, preliminary study which will assess patients prospectively and attempt to correlate markers on genes and single nucleotide polymorphisms with patient phenotypes. This method which will serve as the foundation for a future genome wide association study of pain. This is a preliminary, developmental, prospective follow-up study to develop a tool that will be sensitive and specific enough to be used in a large-scale candidate genome association pain study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Undergoing a primary, unilateral total knee arthroplasty for the first time
* Willing and able to provide informed consent
* Caucasian
* Non-hispanic

Exclusion Criteria:

* Contraindication or refusal for peripheral nerve blocks
* Any chronic pain condition which may confound the study per investigator's opinion
* Chronic opioid dependence per investigator's opinion
* Any diagnosis for total knee arthroplasty other than degenerative joint disease or osteoarthritis
* Evidence of clinical dementia, dementia, delirium, or any cognitive disorder which inhibits the subject's ability to comprehend and cooperate with researchers
* Revision or any knee surgery that is not a primary, unilateral, elective total knee arthroplasty being performed for the first time
* Any criteria that in the investigator's opinion would prohibit the subject from following
* Hispanic ethnicity
* Any race other than caucasian
* Subjects with knee flexion contracture (which is clinically defined for the purpose of our protocol as more than 15 degrees of knee contracture)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04-08 (Actual); Study Completion 2012-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belfer I, Wu T, Kingman A, Krishnaraju RK, Goldman D, Max MB. Candidate gene studies of human pain mechanisms: methods for optimizing choice of polymorphisms and sample size. Anesthesiology. 2004 Jun;100(6):1562-72. doi: 10.1097/00000542-200406000-00032. No abstract available. PMID 15166579
- [Background] Tegeder I, Costigan M, Griffin RS, Abele A, Belfer I, Schmidt H, Ehnert C, Nejim J, Marian C, Scholz J, Wu T, Allchorne A, Diatchenko L, Binshtok AM, Goldman D, Adolph J, Sama S, Atlas SJ, Carlezon WA, Parsegian A, Lotsch J, Fillingim RB, Maixner W, Geisslinger G, Max MB, Woolf CJ. GTP cyclohydrolase and tetrahydrobiopterin regulate pain sensitivity and persistence. Nat Med. 2006 Nov;12(11):1269-77. doi: 10.1038/nm1490. Epub 2006 Oct 22. PMID 17057711
- [Background] Buvanendran A, Kroin JS, Berger RA, Hallab NJ, Saha C, Negrescu C, Moric M, Caicedo MS, Tuman KJ. Upregulation of prostaglandin E2 and interleukins in the central nervous system and peripheral tissue during and after surgery in humans. Anesthesiology. 2006 Mar;104(3):403-10. doi: 10.1097/00000542-200603000-00005. PMID 16508385
- [Background] Tegeder I, Adolph J, Schmidt H, Woolf CJ, Geisslinger G, Lotsch J. Reduced hyperalgesia in homozygous carriers of a GTP cyclohydrolase 1 haplotype. Eur J Pain. 2008 Nov;12(8):1069-77. doi: 10.1016/j.ejpain.2008.02.004. Epub 2008 Apr 18. PMID 18374612
- [Background] Silverman DG, O'Connor TZ, Brull SJ. Integrated assessment of pain scores and rescue morphine use during studies of analgesic efficacy. Anesth Analg. 1993 Jul;77(1):168-70. No abstract available. PMID 8317727
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Reynolds LW, Hoo RK, Brill RJ, North J, Recker DP, Verburg KM. The COX-2 specific inhibitor, valdecoxib, is an effective, opioid-sparing analgesic in patients undergoing total knee arthroplasty. J Pain Symptom Manage. 2003 Feb;25(2):133-41. doi: 10.1016/s0885-3924(02)00637-1. PMID 12590029
- [Background] Max MB, Stewart WF. The molecular epidemiology of pain: a new discipline for drug discovery. Nat Rev Drug Discov. 2008 Aug;7(8):647-58. doi: 10.1038/nrd2595. Epub 2008 Jun 27. PMID 18587382
- [Background] Khan AA, Owatz CB, Schindler WG, Schwartz SA, Keiser K, Hargreaves KM. Measurement of mechanical allodynia and local anesthetic efficacy in patients with irreversible pulpitis and acute periradicular periodontitis. J Endod. 2007 Jul;33(7):796-9. doi: 10.1016/j.joen.2007.01.021. Epub 2007 Mar 26. PMID 17804314
- [Background] Kalff JC, Turler A, Schwarz NT, Schraut WH, Lee KK, Tweardy DJ, Billiar TR, Simmons RL, Bauer AJ. Intra-abdominal activation of a local inflammatory response within the human muscularis externa during laparotomy. Ann Surg. 2003 Mar;237(3):301-15. doi: 10.1097/01.SLA.0000055742.79045.7E. PMID 12616113
- [Background] Gueorguieva RV, Sanacora G. Joint analysis of repeatedly observed continuous and ordinal measures of disease severity. Stat Med. 2006 Apr 30;25(8):1307-22. doi: 10.1002/sim.2270. PMID 16217846
- [Background] Granot M, Ferber SG. The roles of pain catastrophizing and anxiety in the prediction of postoperative pain intensity: a prospective study. Clin J Pain. 2005 Sep-Oct;21(5):439-45. doi: 10.1097/01.ajp.0000135236.12705.2d. PMID 16093750
- [Background] Dionne RA, Berthold CW. Therapeutic uses of non-steroidal anti-inflammatory drugs in dentistry. Crit Rev Oral Biol Med. 2001;12(4):315-30. doi: 10.1177/10454411010120040301. PMID 11603504
- [Background] Dina OA, Hucho T, Yeh J, Malik-Hall M, Reichling DB, Levine JD. Primary afferent second messenger cascades interact with specific integrin subunits in producing inflammatory hyperalgesia. Pain. 2005 May;115(1-2):191-203. doi: 10.1016/j.pain.2005.02.028. PMID 15836982
- [Background] Curatolo M, Petersen-Felix S, Arendt-Nielsen L. Sensory assessment of regional analgesia in humans: a review of methods and applications. Anesthesiology. 2000 Dec;93(6):1517-30. doi: 10.1097/00000542-200012000-00025. No abstract available. PMID 11149448
- [Background] Chan VW, Clark AJ, Davis JC, Wolf RS, Kellstein D, Jayawardene S. The post-operative analgesic efficacy and tolerability of lumiracoxib compared with placebo and naproxen after total knee or hip arthroplasty. Acta Anaesthesiol Scand. 2005 Nov;49(10):1491-500. doi: 10.1111/j.1399-6576.2005.00782.x. PMID 16223396
- [Result] Belfer I, Greco CM, Lokshin A, Vulakovich K, Landsittel D, Dai F, Crossett L, Chelly JE. The design and methods of genetic studies on acute and chronic postoperative pain in patients after total knee replacement. Pain Med. 2014 Sep;15(9):1590-602. doi: 10.1111/pme.12487. Epub 2014 Jul 8. PMID 25040948

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Knee Arthroplasty Subjects Who Are Genotyped
Started | 156
Completed | 153
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Total Knee Arthroplasty Subjects Who Are Genotyped
Number analyzed (Participants) | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 92
  >=65 years | 64
Age, Continuous [Mean (Full Range); unit: years] | 64.23 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 156

OUTCOME MEASURES:

1. Primary Outcome: NRS-Pain With Movement on POD 2
Description: The primary endpoint is the pain reported by subjects, using the NRS-Pain with movement on the second day after surgery.The assumption behind this study is that certain genetic variants (e.g. single-nucleotide polymorphism (SNP) are responsible for part of total variation of certain clinical phenotypes (e.g. post-operative pain here).
  Numeric Rating Score Pain Assessment (0-10 scale where 0 indicates no pain at all and 10 indicates the worst pain imaginable) on Post Op Day 2, Pain with Movement
Time Frame: Postoperative day (POD) 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Total Knee Arthroplasty Subjects Who Are Genotyped
Number analyzed (Participants) | 156
units on a scale | 2.83 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Total Knee Arthroplasty Subjects Who Are Genotyped
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156
Other Adverse Events (participants affected / at risk) | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No